CLINICAL TRIAL: NCT00001101
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial of the Safety and Efficacy of Ceftriaxone and Doxycycline in the Treatment of Patients With Seropositive Chronic Lyme Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMID 97-002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-03

CONDITIONS: Lyme Disease
MeSH Terms: conditions — Lyme Disease | interventions — Ceftriaxone; Doxycycline

INTERVENTIONS:
Drug: ceftriaxone
Drug: doxycycline

SUMMARY:
Lyme disease is the most common tick-borne disease in the United States. It is caused by the spirochete Borrelia burgdorferi. It may exist in a chronic form and be the result of: 1) active infection by B. burgdorferi; 2) damage caused by the original infectious process; or 3) the presence of co-infection with another organism transmitted by Ixodes ticks. The purpose of this study is to determine the safety and effectiveness, for seropositive patients, of intensive antibiotic treatment in eliminating symptoms of Chronic Lyme Disease (CLD).

DETAILED DESCRIPTION:
One hundred ninety-four (194) patients will be enrolled in this study. Each patient will be assigned to one of two groups and will be randomly selected to receive either antibiotic therapy or placebo; but, the assignment of medication will not be made known to the patient or administering doctor. Antibiotic or placebo will be given intravenously (IV) for 30 consecutive days and then orally for the next 60 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Are 18 years of age or older.
* Are seropositive for antibodies against B. burgdorferi antigens by Western Blot at enrollment.
* Have documented history of acute Lyme disease.
* Have had a rash (erythema migrans) that resembles a bullseye. This skin aberration usually occurs after a tick bite in late spring, summer or early fall and is sometimes accompanied by fatigue, fever, headache, mild stiff neck, arthralgia or myalgia.
* Have had one or more clinical features typical of Lyme disease acquired in the United States (see technical summary).
* Have had one or more of the following symptoms and conditions that have persisted for at least 6 months (but less than 12 years) and are not attributable to another cause or condition: a) widespread musculoskeletal pain and fatigue that began coincident with or within 6 months following initial infection with B. burgdorferi. b) certain neurologic symptoms including memory impairment and nerve pain within 6 months following initial infection with B. burgdorferi.
* Have had a physician-documented history of prior antibiotic treatment with a currently recommended antibiotic regimen.

Exclusion Criteria:

You will not be eligible for this study if you:

* Have previously enrolled in this study.
* Are pregnant, lactating, or unable to use birth control measures during the treatment period of this study.
* Are taking chronic medication that could interfere with evaluation of symptoms.
* Are taking or have taken various medications that could interfere with the evaluation of symptoms (see technical summary).
* Are hypersensitive to ceftriaxone or doxycycline.
* Have active inflammatory synovitis.
* Have another disease that could account for symptoms of acute Lyme disease.
* Have another serious disease or an active infection.
* Are unable to tolerate an IV.
* Have tested positive for Borrelia DNA in plasma or cerebrospinal fluid at the time of initial evaluation for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194
Dates: Primary Completion 2001-03 (Actual); Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mark Klempner, Boston, Massachusetts, United States

REFERENCES:
- [Background] Klempner MS, Hu LT, Evans J, Schmid CH, Johnson GM, Trevino RP, Norton D, Levy L, Wall D, McCall J, Kosinski M, Weinstein A. Two controlled trials of antibiotic treatment in patients with persistent symptoms and a history of Lyme disease. N Engl J Med. 2001 Jul 12;345(2):85-92. doi: 10.1056/NEJM200107123450202. PMID 11450676
- [Background] Klempner MS, Schmid CH, Hu L, Steere AC, Johnson G, McCloud B, Noring R, Weinstein A. Intralaboratory reliability of serologic and urine testing for Lyme disease. Am J Med. 2001 Feb 15;110(3):217-9. doi: 10.1016/s0002-9343(00)00701-4. No abstract available. PMID 11182109
- [Background] Perides G, Charness ME, Tanner LM, Peter O, Satz N, Steere AC, Klempner MS. Matrix metalloproteinases in the cerebrospinal fluid of patients with Lyme neuroborreliosis. J Infect Dis. 1998 Feb;177(2):401-8. doi: 10.1086/514198. PMID 9466528
- [Background] Klempner M, Hu L, Johnson G. Severe physical disability and other characteristics in patients with post treatment chronic Lyme disease. VIII International Conference on Lyme Borreliosis and other Emerging Tick-Borne Diseases, Munich, Germany June 20-24, 1999.